CLINICAL TRIAL: NCT07381491
Title: Effects of Core Strengthening With Pelvic Proprioceptive Neuromuscular Facilitation on Trunk Control and Balance in Patients With Sub-acute Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/21686
Record Dates: First submitted 2025-12-23; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: Stroke; PNF; Core Strengthening; Trunk control; Balance Impairment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Masking Description: This single-blind randomized controlled study evaluated the effectiveness of core stabilization combined with pelvic PNF on trunk control and balance in post-stroke individuals. Participants were blinded to group allocation to reduce expectation bias, while therapists and assessors were unblinded due to intervention requirements. The study aimed to address a gap in evidence regarding this combined approach and to support evidence-based stroke rehabilitation practices that enhance trunk function, balance, and functional independence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants who were included in this group got Pelvic Proprioceptive neuromuscular facilitation techniques + core strengthening group + Trunk control exercises (Conventional treatment).
  Interventions: Other: Core stabilization exercises; Other: PNF; Other: Trunk control exercises
- Control Group (Other): Participants in group 2 received Core stabilization exercises + Conventional trunk control exercises (Rhythmic stabilization, Bridging, Side-Lying Trunk Lifts, Quadruped, Kneeling and modified plantigrade positioning) exercises. 3 sets with 10 repetitions each, 3 sec rest between each repetition, 1 min rest after each set and 3 min rest between each exercise.
  Interventions: Other: Core stabilization exercises; Other: Trunk control exercises

INTERVENTIONS:
Other: Core stabilization exercises — Core activated by Bio Feedback apparatus and participants were given instructions to do trunk curls in crook lying position. Asked to lift their upper trunk slightly (15 degree) from the plinth. 3 sets with 10 repetitions each, 3 sec rest between each repetition, 1 min rest after each set and 3 min rest between each exercise.
Other: PNF — Proprioceptive neuromuscular facilitation techniques The sequence was rhythmic initiation, slow reversal then agonistic reversals. each technique was applied for 3 sets of 2 min duration each with 30 sec between each set and 2 min rest after each technique. A stopwatch was used to measure the time.
  Arms: Experimental Group
Other: Trunk control exercises — Trunk control exercises Different trunk exercises were performed by the participants to develop trunk control and balance. Rhythmic stabilization, Side-Lying Trunk Lifts, Bridging, Quadruped, Kneeling and modified plantigrade positioning, are the trunk exercises which were used conventionally to develop trunk control. 3 sets with 10 repetitions each, 3 sec rest between each repetition, 1 min rest after each set and 3 min rest between each exercise.

SUMMARY:
Purpose of this study was to investigate the effectiveness of core stabilization with pelvic proprioceptive neuromuscular facilitation on trunk control and balance which will be provided an evidence-based selection of the best possible intervention to improve trunk function and balance as compared to the trunk control exercises such as Rhythmic stabilization, Bridging, Side-Lying Trunk Lifts, Quadruped, Kneeling and modified plantigrade positioning, which one can provide the better balance and trunk control in sub-acute stroke patients.

DETAILED DESCRIPTION:
Interventions FITT Principle Intervention was given for 60 min per session (30 + 30 mins for each group), including 3 sets with10 repetitions each, 3 sec rest between each repetition, 1 min rest after each set and 3 min rest between each exercise (this FITT principle for core stabilization and trunk control exercises). For PNF technique each technique was applied for 3 sets of 2 min duration each with 30 sec between each set and 2 min rest after each technique.

Once a day, 5 times per week for 6 weeks for both groups. Groups There were two groups Groups 1 (interventional group) Groups 2 (control group) Groups 1 (interventional group) Participants who were included in this group got Pelvic Proprioceptive neuromuscular facilitation techniques + core strengthening group + Trunk control exercises (Conventional treatment).

Core stabilization exercises techniques Core activated by Bio Feedback apparatus and participants were given instructions to do trunk curls in crook lying position. Asked to lift their upper trunk slightly (15 degree) from the plinth. 3 sets with 10 repetitions each, 3 sec rest between each repetition, 1 min rest after each set and 3 min rest between each exercise.

Proprioceptive neuromuscular facilitation techniques The sequence was rhythmic initiation, slow reversal then agonistic reversals. each technique was applied for 3 sets of 2 min duration each with 30 sec between each set and 2 min rest after each technique. A stopwatch was used to measure the time.

Trunk control exercises Different trunk exercises were performed by the participants to develop trunk control and balance. Rhythmic stabilization, Side-Lying Trunk Lifts, Bridging, Quadruped, Kneeling and modified plantigrade positioning, are the trunk exercises which were used conventionally to develop trunk control. 3 sets with 10 repetitions each, 3 sec rest between each repetition, 1 min rest after each set and 3 min rest between each exercise.

Groups 2 (control group) Participants in group 2 received Core stabilization exercises + Conventional trunk control exercises (Rhythmic stabilization, Bridging, Side-Lying Trunk Lifts, Quadruped, Kneeling and modified plantigrade positioning) exercises. 3 sets with 10 repetitions each, 3 sec rest between each repetition, 1 min rest after each set and 3 min rest between each exercise.

Core stabilization exercises techniques Core activated by Bio Feedback apparatus and participants were given instructions to do trunk curls in crook lying position. Asked to lift their upper trunk slightly (15 degree) from the plinth. 3 sets with 10 repetitions each, 3 sec rest between each repetition, 1 min rest after each set and 3 min rest between each exercise.

Trunk control exercises Different trunk exercises were performed by the participants to develop trunk control and balance. Rhythmic stabilization, Side-Lying Trunk Lifts, Bridging, Quadruped, Kneeling and modified plantigrade positioning, are the trunk exercises which were used conventionally to develop trunk control. 3 sets with 10 repetitions each, 3 sec rest between each repetition, 1 min rest after each set and 3 min rest between each exercise.

Outcomes Measures Trunk Impairment Scale (TIS) is a standardized scale to assess the trunk function and stability in stroke patients(39). We used the pre- and post-intervention scores of Trunk Impairment Scale (TIS) to evaluate trunk function and stability.

Berg Balance Scale (BBS) is identified as the most commonly used as an evaluation tool in the stroke rehabilitation(40). We used the pre- and post-intervention scores of Berg Balance Scale (BBS) to evaluate the balance.

Data Collection Procedure The study was conducted by informed consent from participants. Assessment was performed before the intervention and after the intervention (after 6 weeks) from Trunk Impairment Scale (TIS) and Berg Balance Scale (BBS). Pre-interventional and post interventional scores were documented and analyzed the according to the statistical method.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 45 and 60 years.
* Sub-acute phase of unilateral ischemic stroke.
* More than two weeks but no more than six months were included.
* Participants should be able to walk with or without support for 2-4 min.
* Participants with modified Ashworth scale grade 1 or grade 2.
* Participants should be able to understand and follow simple verbal instructions (Mini-Mental Status Examination [MMSE]≥24).

Exclusion Criteria:

* Participants with recurrent stroke; brainstem or cerebellar stroke or hemorrhagic stroke.
* Participants with modified Ashworth scale grade ≥3 (severe spasticity).

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Trunk Impairment Scale | • Baseline • After 6 weeks
  The Trunk Impairment Scale (TIS) is a 17-item clinical tool assessing stroke patients across three subscales-static sitting balance (0-7 points), dynamic sitting balance (0--10points), and trunk coordination (0-6 points)-totaling a maximum score of 23. Higher scores indicate better, more controlled, and coordinated trunk function, with evaluations performed in a seated position.
Berg Balance Scale | • Baseline • After 6 weeks
  Berg Balance Scale (BBS) is identified as the most commonly used as an evaluation tool in the stroke rehabilitation. We used the pre- and post-intervention scores of Berg Balance Scale (BBS) to evaluate the balance. Total score of berg balance scale is 56.Highest score shows the low fall risk and the lowest score shows the high fall risk.

CONTACTS AND LOCATIONS:
Overall Officials: NABEELA Dawood, Study Chair — Lahore University of Biological and Applied Sciences
Locations (1):
- Ghurki Trust & Teaching Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No